CLINICAL TRIAL: NCT04913441
Title: Effects of Manual Therapy Versus Stretching Versus Routine Physical Therapy on Pain, ROM, and Functional Disability in Restaurant Chef Workers With Nonspecific Chronic Neck Pain: A Randomised Controlled Trial
Brief Title: Manual Therapy vs Stretching vs Routine Physical Therapy in Nonspecific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS/FSD/REC/0260
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Neck Pain
Keywords: Neck pain; Manual therapy; Stretching exercises; Physical Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study would be double blinded as accessor and the participant of the study would be kept blind of the treatment group to which patient would be allocated. After the complete initial screening process, every recruited patient will be accessed by an independent assessor, expert will use outcome measuring tools. his will be recorded as baseline measurement assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine physical therapy (Experimental): Patients in this group will get every session of 30 min 3 times per week on alternative days for 12 weeks
  1. TENS and hot pack for 15 minutes
  2. Ultra sound for 5 minutes
  3. ROM exercises repeats 5 times for 10 minutes
  Interventions: Other: Routine physical therapy
- Manual physical therapy with routine physical therapy (Experimental): Patients in group B will get every session 30 minutes 3 times per week on alternative days
  1. TENS and hot pack for 15 minutes
  2. Ultra sound for 5 minutes
  3. Mulligan technique (NAGS and SNAGS) will repeats 5 times for 10 minutes
  Interventions: Other: Manual physical therapy with routine physical therapy
- Stretching physical therapy with routine physical therapy (Experimental): Patients in this group will get every session 30 minutes 3 times per week on alternative days
  1. TENS and hot pack for 15 minutes
  2. Ultra sound for 5 minutes
  3. Stretching exercises repeats 5 times for 10 minutes
  Interventions: Other: Stretching physical therapy with routine physical therapy

INTERVENTIONS:
Other: Routine physical therapy — Patients in this group will get every session routine physical therapy of 30 minutes 3 times per week on alternative days for 12 weeks
  Other Names: Rehabilitation following Routine physical therapy
  Arms: Routine physical therapy
Other: Manual physical therapy with routine physical therapy — Patients in this group will get every session Manual physical therapy with routine physical therapy of 40 to 45 minutes 3 times per week on alternative days for 12 weeks
  Other Names: Rehabilitation following Manual physical therapy with routine physical therapy
  Arms: Manual physical therapy with routine physical therapy
Other: Stretching physical therapy with routine physical therapy — Patients in this group will get every session of Stretching physical therapy with routine physical therapy of 40 to 45 minutes 3 times per week on alternative days for 12 weeks
  Other Names: Rehabilitation following Stretching physical therapy with routine physical therapy
  Arms: Stretching physical therapy with routine physical therapy

SUMMARY:
The aim of this study is to analyze the effect of Mulligan technique vs stretching techniques and vs routine physical therapy on pain ,range of motion(ROM) and functional disability among restaurant chefs with non-specific chronic pain.

DETAILED DESCRIPTION:
Neck pain (NP) is one of the basic musculoskeletal issues. Neck pain can be due to stress about the musculoskeletal framework because of postural problems and may be related with different causes, such as: - Intervertebral disc herniation, -nerve compression -fracture.

Nonspecific neck pain is a pain located in the lateral and posterior neck that does not show pathognomonic signs and symptoms. When the duration of symptoms is greater than 12 weeks of evolution, it acquires the value of chronicity, being denominated non-specific chronic neck pain (NCNP). It is a common disorder, which generates a great impact and socio-economic cost .

In this study we evaluate the comparison of manual physical therapy vs routine physical therapy vs stretching physical therapy effects among restaurants chefs having non-specific chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain for atleast 3 months having no :

  * Neurological Problem
  * Rheumatological Problem
  * Patient had taken any analgesic medication for neck pain for last 3 months.
  * Non specific neck pain
  * Age 18-60 years

Exclusion Criteria:

* Neck pain due to,

  * Tumors
  * Ankylosings Spondylitis
  * Fracture
  * Dislocation
  * Presence of cord compression
  * Vertebrobasilar artery insufficiency
  * Osteoprosis OR Osteopenia
  * Long term use of anticoagulant or corticosteroid drugs
  * Pain due to any congenital deformity, inflammation or any infection
  * Carcinoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | 3 months
  Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain
Bubble inclinometer | 3 months
  Baseline's Bubble Inclinometer is a simple to use device for measuring range of motion in patients. The inclinometer can be used to measure range of motion in the neck, the hip, the elbow, the knee, the shoulder, the spine, the ankle, the wrist, and the MCP joint

SECONDARY OUTCOMES:
Neck disability Index (NDI) | 3 months
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No